CLINICAL TRIAL: NCT04828655
Title: Análisis de Medidas bioparamétricas Para Correlacionar Los hábitos Diarios y Reducir la tensión Arterial
Brief Title: Analysis of Bioparametric Measures for Correlating Daily Habits and Reducing Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Assistant Professor, University of Alicante
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: UA-2020-04-16
Record Dates: First submitted 2021-03-23; First posted 2021-04-02 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Hypertension; Diet, Mediterranean; Cardiovascular Diseases; Exercise; Machine Learning; Overweight and Obesity; Body Composition; Triglyceride-Storage; Disease
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Motor Activity; Overweight; Obesity; Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): Recommendations on healthy eating habits based on the Mediterranean diet and moderate physical activity. Specific micronutrient intake focused on improving cardiovascular parameters and body composition.
- EXPERIMENTAL GROUP (Experimental): Recommendations on healthy eating habits based on the Mediterranean diet and moderate physical activity through an application based on machine learning. Intake of specific micronutrients focused on improving cardiovascular parameters and body composition.
  Interventions: Behavioral: Use of a mobile application based on machine learning with the aim of improving health and body composition parameters.

INTERVENTIONS:
Behavioral: Use of a mobile application based on machine learning with the aim of improving health and body composition parameters. — Specific diet program and moderate physical activity, all guided and mediated by a mobile application. As well as the recording and monitoring of periodic evaluations of health indicators.
  Arms: EXPERIMENTAL GROUP

SUMMARY:
To study the effects of the use of a mobile application plus recommendations based on a Mediterranean diet on the intake of micronutrients from natural sources (not drugs) on health indicators, cardiovascular parameters (blood pressure...), physical condition and body composition in a Spanish adult population.

DETAILED DESCRIPTION:
In the Valencian Community, 93% of deaths appear to be related to (non-communicable) diseases such as: obesity, hypertension and diabetes. In 2013, cardiovascular diseases were the leading cause of death in women (34.4%) and the second in men (28.0%). There is a forecast that overweight and obesity will reach levels of 89% and 85% in men and women, respectively, by 2030. This will result in an increase in the obesity-related prevalence of coronary heart disease by 97%. The promotion of research on arterial hypertension and how it could be reduced is one of the basic pillars in decreasing the prevalence and incidence in the Spanish population. Research should anticipate and develop treatments and vaccines that prevent new scenarios of widespread infection.

Therefore, the main objective is to study the effects of the use of a mobile application plus recommendations based on a Mediterranean diet on the intake of micronutrients from natural sources (not drugs) on health indicators, cardiovascular parameters (blood pressure...), physical condition and body composition in the adult Spanish population.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years old
* Healthy.
* Blood pressure levels slightly elevated but less than 140 mm Hg and/or diastolic pressure less than 90 mm Hg.
* Smartphone access

Exclusion Criteria:

* Subjects with diseases.
* Consumption of drugs and/or supplements.
* Subjects with food intolerances/allergies.
* Subjects with muscle or joint injury.
* Subjects with impossibility to follow up the intervention.
* Refusal of informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiovascular variables; heart rate. | 9 months
  Heart rate measurement done with an activity wristband.
Cardiovascular variables; blood pressure. | 9 months
  Measurement of blood pressure (systolic and diastolic) with a digital tensiometer.
Physical condition; time. | 9 months
  The evaluation of the physical condition will be carried out by means of the mile test, in which the subjects have to cover this distance walking, and in the shortest possible time.
Body Composition - Bioimpedance | 9 months
  Assessment of body composition using the TANITA (Tokyo, Japan) validated bioimpedance scale to obtain the results of fat mass, fat-free mass and visceral mass.
Weight | 9 months
  The weight of the subjects will be obtained using the TANITA (Tokyo, Japan). From the body mass and height data, the BMI (kg/m2) will be obtained.
Height | 9 months
  The height of the subjects will be measured with the SECA 123 stadiometer (Hamburg, Germany). From the body mass and height data, the BMI (kg/m2) will be obtained.
Body Composition - Skinfolds | 9 months
  The kinanthropometric assessment will be carried out using the methodology proposed for the restricted profile by the International Society for the Development of Kineanthropometry (ISAK). The material used to measure skinfolds will be a plicometer.
Body Composition - Perimeters | 9 months
  The kinanthropometric assessment will be carried out using the methodology proposed for the restricted profile by the International Society for the Development of Kineanthropometry (ISAK). The material used to measure perimeters will be a tape.
Body Composition - Diameters | 9 months
  The kinanthropometric assessment will be carried out using the methodology proposed for the restricted profile by the International Society for the Development of Kineanthropometry (ISAK). The material used to measure diameters will be a pachymeter.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Martínez Rodríguez, Principal Investigator — Alicante University
Locations (1):
- Alejandro Martínez Rodriguez, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No